CLINICAL TRIAL: NCT06463262
Title: Exploration of Personalized Biomarkers During Neoadjuvant Radiation Therapy for Spinal and Sacral Chordoma
Acronym: Canon
Status: Recruiting | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: J2317; IRB00291203 (Other: JHM IRB)
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Chordoma of Spine; Chordoma of Skull Base; Chordoma of Sacrum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal, Sacral Chordoma
  Interventions: Diagnostic Test: ctDNA

INTERVENTIONS:
Diagnostic Test: ctDNA — the effects of neoadjuvant RT, in the form of either proton therapy or SBRT, on the ctDNA

SUMMARY:
In this study the investigators will study the effects of neoadjuvant radiation therapy (RT), in the form of either proton therapy or stereotactic body radiation therapy (SBRT), on the Circulating tumor DNA (ctDNA), radiographic changes and radiomics, and the validity of these findings will be compared using the current gold standard- pathologic findings. The purpose of this work is to explore whether the biomarkers may be used diagnostically to better understand radiographic changes following RT. The investigators hypothesize that ctDNA levels in combination with imaging biomarkers identified through radiomics will be a sensitive and specific tool for predicting histopathologic response to RT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically proven chordoma of the skull base, spine, or sacrum (coccyx lesions are eligible).
* Radiographic evidence of spinal sacral chordoma is required and may be obtained from computed tomography imaging and/or magnetic resonance imaging. Other studies may be used with principal investigator approval.

Note: Patients enrolled in Dr. Chetan Bettegowda's J1576 study, (IRB00075499) may be considered eligible for this trial. The J1576 study enrolls patients who have been diagnosed with Chordoma. Prior to enrollment, all patients must be consented specifically for participation in this Chordoma study (IRB00291203).

* Treating physician must deem that neoadjuvant proton therapy or SBRT is appropriate treatment for the chordoma.
* Surgical resection with curative intent must be planned.
* The patient must have a Karnofsky Performance Score of 40 or greater.
* If a woman is of child-bearing potential, a negative urine or serum pregnancy test must be demonstrated prior to treatment. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for up to 12 weeks following the study. Should a woman become pregnant or suspect she is pregnant while participating in this study she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior radiation or radiosurgery to the involved level of the spine.
* Patients with metastatic disease will be excluded.
* Prior malignancies are excluded except for adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, or other cancer from which the patient has been disease free for at least 1 year.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements will be excluded.
* Pregnant women are excluded. Women of child-bearing potential who are unwilling or unable to use and acceptable method of birth control to avoid pregnancy for the entire study period and up to 12 weeks after the study are excluded. Male subjects must also agree to use effective contraception for the same period as above.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Potential participants who are clinical patients of the PI or co-investigators may be identified during chart review in advance of a routine clinic visit or during a routine clinic visit with a provider.
  Patients who are enrolled in IRB: IRB00075499 (PI: Dr. Chetan Bettagowda) may be eligible for this trial as well. Once identified as a potential study participant, the study team for this ctDNA study would have to confirm eligibility as for any potential participant.
  In addition, potential participants may contact the study team directly.
  Some of these potential participants may also be identified during the multidisciplinary clinic as part of the standard clinic case review process.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of combining ctDNA and radiomics | within one week after surgery
  Sensitivity and specificity of combining ctDNA and radiomic features in predicting histopathologic changes at surgery defined by patients who have <10% necrosis, the percentage of patients who are deemed "positive" by the model based on ctDNA and radiomics

SECONDARY OUTCOMES:
Percent of necrotic and active tumor cells | within one week after surgery
  Percent of necrotic and active tumor cells following neoadjuvant RT using proton therapy or SBRT according to the Johns Hopkins Solid Tumor Panel Next Generation Sequencing
Change in plasma ctDNA levels | within one week after surgery
  Change in plasma ctDNA levels following neoadjuvant RT for spinal chordoma and correlate changes in ctDNA levels with histopathologic changes at surgery
Correlate radiomic features with histopathologic and genomic features | within one week after surgery
  Correlate radiomic features with histopathologic and genomic features in patients receiving neoadjuvant RT for spinal and sacral chordoma
Radiographic local recurrence | within one week after surgery
  Radiographic local recurrence defined as evidence of progressive disease on CT/MRI in the operative site when compared to post-op imaging.
Rate of wound healing complications | within one week after surgery
  Rate of wound healing complications following neoadjuvant RT for spinal chordoma
Health related quality of life as assessed by the European Organization for Research and Treatment of Cancer (EORTC) quality of life (QLQ-C15-PAL) questionnaire | within one week after surgery
  Health related quality of life following neoadjuvant RT for spinal chordoma measured by the European Organization for Research and Treatment of Cancer (EORTC) quality of life (QLQ-C15-PAL) questionnaire. The scoring ranges from 0-21, with 21 being the highest quality of life.
Local progression free survival | 3 years
  Local progression free survival following neoadjuvant RT for spinal chordoma
Overall survival | 3 years
  Overall survival following neoadjuvant RT for spinal chordoma
Relationship between ctDNA post-op and local Progression Free Survival (PFS) | 3 years
  The relationship between circulating tumor DNA post-operatively and local PFS following neoadjuvant RT for spinal chordoma
Relationship between ctDNA post-op and Overall Survival (OS) | 3 years
  The relationship between circulating tumor DNA post-operatively and OS following neoadjuvant RT for spinal chordoma
Toxicity of neoadjuvant RT as assessed by CTCAE version 5 | 3 years
  Toxicity of neoadjuvant RT for chordoma using CTCAE version 5

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Redmond, MD, MPH, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania